CLINICAL TRIAL: NCT01877564
Title: A Randomized Pilot Study to Evaluate the Effects of a Short Course of Metformin Versus No Therapy in the Period Prior to Hysterectomy for Grade 1-2 Adenocarcinoma of the Endometrium in Obese Non-Diabetic Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 138647
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Adenocarcinoma of the Endometrium
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Metformin (Experimental): oral metformin at 500 mg twice a day for 14-21 days followed by surgery
  Interventions: Drug: Metformin
- Group 2 - No treatment (No Intervention)

INTERVENTIONS:
Drug: Metformin
  Arms: Group 1 - Metformin

SUMMARY:
The purpose of this research is to determine the effects of Metformin, a well tolerated drug widely prescribed for treatment of Type 2 Diabetes Mellitus, on endometrium cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed diagnosis of grade I or II adenocarcinoma of the endometrium
* Must be obese as defined by a body mass index (BMI) greater than or equal to 30 kg/m2
* Candidate for surgical removal of their uterus as part of their endometrial cancer treatment
* Subjects must have signed informed consent
* Age 42 - 65 years of age
* Electrocorticogram (ECOG) Performance status of 0 - 2
* History of adequate renal, liver, and bone marrow function:

  * Hb: (adequate for surgical intervention, with transfusion if necessary) White Blood Cell (WBC): (normal range)
  * Platelets: (180K/cmm)
  * Liver Function Test(LFTs): Normal bilirubin (<2.0mg/dL), AST/ALT (2xULN)
  * Renal function: creatinine less than 1.4
* Female subjects must either not be of child-bearing potential or must have a negative urine pregnancy test within 7 days of randomization to Metformin. Subjects are considered not of child-bearing potential if they are surgically sterile or they are postmenopausal for greater than 12 months.

Exclusion Criteria:

* Poorly differentiated cancer or any of the high-risk subtypes of endometrial cancer including serous, clear cell, or carcinosarcoma
* History of diabetes mellitus Type 1 or Type 2.
* Receiving metformin prior to enrollment
* Known hypersensitivity to metformin.
* Unable to swallow and retain oral medication.
* Pregnant or lactating.
* Previous or concurrent malignancies, except non-melanoma skin cancers, unless curatively treated and with no evidence of recurrence for > 5 years
* If the physician feels that the candidate is not suitable for the study, he/she will be excluded.
* Currently taking biguanides, sulfonylurea drugs, thiazolidinediones, insulin, or mTOR or DPP-4 inhibitors or having taken any of these medications during the 12 weeks prior to study participation.
* Clinical symptoms of gastrointestinal obstruction or bleeding and consideration for immediate surgery or immediate neoadjuvant chemoradiation.
* History of lactic or other metabolic acidosis.
* Uncontrolled infectious disease.
* History of positivity for human immunodeficiency virus (HIV).
* History of congestive heart failure requiring pharmacologic treatment.
* History of excessive alcohol abuse, defined by a habitual intake of more than three drinks daily.
* Mal-absorption syndrome, disease affecting gastrointestinal function, or previous resection of the stomach or small bowel.
* Current use of medications for weight loss.
* Currently taking cimetidine, thiazide diuretics or cephalexin. If a patient needs some of these agents, alternative agents should be substituted.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2017-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the UAMS Gynecologic Oncology Clinic between August 2013 and July 2016.
Pre-assignment Details: Subject eligibility was established before treatment randomization and included eligibility assessments, study assessments, lab tests, and pathology assessments.
Groups:
- Group 1 - Metformin: oral metformin at 500 mg twice a day for 14-21 days followed by surgery
  Metformin
- Group 2 - No Treatment: no metformin for 14-21 days
Period: Overall Study
Arm/Group | Group 1 - Metformin | Group 2 - No Treatment
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Metformin | Group 2 - No Treatment | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Full Range); unit: years] | 60.6 [42 to 72] | 61 [58 to 63] | 60.8 [42 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: IHC-based Tissue Markers of Proliferation
Time Frame: 1 year
Population: data were not collected
Arm/Group | Group 1 - Metformin | Group 2 - No Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group 1 - Metformin | Group 2 - No Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 1/6 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Metformin (N=6) | Group 2 - No Treatment (N=4)
dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) — painful urination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT01877564/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT01877564/SAP_001.pdf